CLINICAL TRIAL: NCT00796718
Title: An Open Label Study of the Effect of Xeloda and Radiotherapy on Pathological Response Rate in Patients With Locally Advanced Rectal Cancer
Brief Title: A Study of Xeloda (Capecitabine) Plus Radiotherapy in Participants With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21800; 2008-003980-38
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

ARMS (1):
- Capecitabine (Experimental): Capecitabine orally twice daily plus standard radiotherapy for 5 weeks, followed by surgery within 6 weeks after completion of treatment.
  Interventions: Radiation: Standard radiotherapy; Drug: Capecitabine [Xeloda]

INTERVENTIONS:
Radiation: Standard radiotherapy — Administered as prescribed according to normal clinical practice.
Drug: Capecitabine [Xeloda] — 825 milligrams per meter square (mg/m^2) orally twice daily for 5 weeks.
  Other Names: Xeloda®

SUMMARY:
This single arm study will assess the efficacy and safety of treatment with Xeloda plus standard pelvic radiotherapy in participants with locally advanced rectal cancer. Eligible participants will receive Xeloda 825mg/m^2 orally twice daily plus standard radiotherapy for 5 weeks, followed by surgery within 6 weeks after completion of treatment. The anticipated time on study treatment is < 3 months, and the target sample size is < 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-80 years of age;
* rectal cancer;
* planned surgery, and likely to benefit from pre-operative combined chemo-radiotherapy;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* previous radiotherapy or chemotherapy for colorectal cancer;
* clinically significant cardiovascular disease;
* significant gastric or small intestine disease;
* serious uncontrolled active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Slovakia (2):
  - Banská Bystrica
  - Bratislava

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 62 participants were enrolled in the study.
Groups:
- Capecitabine: Capecitabine 825 milligrams per meter square (mg/m^2) orally twice daily plus standard radiotherapy for 5 weeks as prescribed according to normal clinical practice, followed by surgery within 6 weeks after completion of treatment.
Period: Overall Study
Arm/Group | Capecitabine
Started | 62
Completed | 53
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Exclusion Criteria | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Informed Consent | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Capecitabine: Capecitabine 825 mg/m^2 orally twice daily plus standard radiotherapy for 5 weeks as prescribed according to normal clinical practice, followed by surgery within 6 weeks after completion of treatment.
Arm/Group | Capecitabine
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response
Description: Pathological complete response was defined as the absence of viable tumor cells in the tumor specimen, including regional lymph nodes determined with standard histological procedures.
Time Frame: Up to 11 weeks (assessed at the time of post-treatment surgery)
Population: Participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 50
percentage of participants | 16

2. Secondary Outcome: Percentage of Participants With Response to Treatment Assessed 4-6 Weeks After the Completion of Radiochemotherapy (Complete Response, Partial Remission or No Response to the Treatment)
Description: Complete response was defined as the disappearance of all target and non-target lesions. Partial remission was defined as ≥ 30% decrease in the sum of the longest diameter (SLD) of target lesions, taking as reference the baseline SLD, or the persistence of 1 or more non-target lesions. No response to treatment was defined as neither sufficient shrinkage to qualify for partial remission nor sufficient increase to qualify for progressive disease, compared to the baseline SLD.
Time Frame: Up to 11 weeks (assessed 4-6 weeks after the completion of radiochemotherapy)
Population: Participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 49
percentage of participants
  Complete Response | 2
  Partial Remission | 12.2
  No Response | 77.6

3. Secondary Outcome: Percentage of Participants With Response to the Treatment Assessed 1 Month After Surgery (Complete Response, Partial Remission or No Response to the Treatment)
Description: as for outcome 2
Time Frame: Up to 15 weeks (assessed 1 month after surgery)
Population: Participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 50
percentage of participants
  Complete Response | 56
  Partial Remission | 10
  No Response | 14

4. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event was defined as any untoward medical occurrence in a participant administered the investigational product which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 15 weeks
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 62
percentage of participants | 91.9

ADVERSE EVENTS:
Time Frame: Up to 15 weeks
Description: All enrolled participants.
Arm/Group | Capecitabine
Serious Adverse Events (participants affected / at risk) | 4/62
Other Adverse Events (participants affected / at risk) | 49/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=62)
Ventricular fibrillation (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Hemorrhoidal inflammation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=62)
Anemia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 7
Rectal pain (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 6
Upper respiratory infection (Infections and infestations) | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 20
Cyst in the liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Erythema (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.